CLINICAL TRIAL: NCT07209826
Title: In Vivo Evaluation of the Scanning Accuracy of Scanners Operating With Different Scanning Technologies in Mandibular and Maxillary Edentulous Ridges
Brief Title: Evaluation of the Scanning Accuracy of Scanners Operating With Different Scanning Technologies in Mandibular and Maxillary Edentulous Ridges
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ayşe Sule NAZLIGUL, Research Assistant, Ege University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Ege-DHF-ASN-01
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-04

CONDITIONS: Accuracy; Measurement Reliability
Keywords: intra-oral scanner; digital impression; Complete Edentulism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Trios 5 Intra-oral scanner (Experimental): It is an intraoral scanner that works with confocal microscopy scanning technology. The purpose of using the intraoral scanner in our work is to take intraoral digital measurements by scanning edentulous ridges. They record the patient's intraoral images in high resolution.
  Interventions: Other: iTero Lumina; Other: Medit i700; Other: E4 Lab Scanner
- Medit i700 Intra-oral Scanner (Experimental): It is an intraoral scanner that works with active triangulation scanning technology. In our study, the purpose of using the intraoral scanner is to take intraoral digital measurements by scanning edentulous ridges. They record the patient's intraoral images in high resolution.
  Interventions: Other: Trios 5; Other: iTero Lumina; Other: E4 Lab Scanner
- iTero Lumina Intra-oral Scanner (Experimental): It is an intraoral scanner that works with multi-unit-capture scanning technology. In this study, using the new generation digital scanning technology of iTero Lumina, intraoral digital measurements are taken by scanning edentulous ridges. They record the patient's intraoral images in high resolution.
  Interventions: Other: Trios 5; Other: Medit i700; Other: E4 Lab Scanner
- E4 Lab Scanner Extra-oral Scanner (Active Comparator): The 3Shape E4 laboratory scanner (EOS) is a desktop laboratory scanner with an indirect scanning procedure. It features fast and accurate scanning technology. With 3Shape E4 scanners, the scanning process begins as soon as you place the model inside the scanner. It records the digital measurement data of the model.
  In our study, the primary model (reference scan) obtained by taking conventional measurements from the patient is scanned using a laboratory scanner, and digital data is obtained.
  Interventions: Other: Trios 5; Other: iTero Lumina; Other: Medit i700

INTERVENTIONS:
Other: Trios 5 — Each patient's edentulous ridges are planned to be scanned three times with Trios 5.To ensure optimum accuracy, scans were performed in a standard dark environment in accordance with the manufacturer's scanning protocols.
  Arms: E4 Lab Scanner Extra-oral Scanner; Medit i700 Intra-oral Scanner; iTero Lumina Intra-oral Scanner
Other: iTero Lumina — Each patient's edentulous ridges are planned to be scanned three times with iTero Lumina.To ensure optimum accuracy, scans were performed in a standard dark environment in accordance with the manufacturer's scanning protocols.
  Arms: E4 Lab Scanner Extra-oral Scanner; Medit i700 Intra-oral Scanner; Trios 5 Intra-oral scanner
Other: Medit i700 — Each patient's edentulous ridges are planned to be scanned three times with Medit i700.To ensure optimum accuracy, scans were performed in a standard dark environment in accordance with the manufacturer's scanning protocols.
  Arms: E4 Lab Scanner Extra-oral Scanner; Trios 5 Intra-oral scanner; iTero Lumina Intra-oral Scanner
Other: E4 Lab Scanner — Conventional measurements will be taken from each patient, and the resulting master model (reference scan) will be scanned using an industrial scanner with high scanning accuracy (E4 lab scanner, 3shape, Denmark) to obtain digital data.
  Arms: Medit i700 Intra-oral Scanner; Trios 5 Intra-oral scanner; iTero Lumina Intra-oral Scanner

SUMMARY:
This study aims to evaluate the scanning accuracy of scanners equipped with Active Triangulation, Confocal Microscopy, and Multi-Direct-Capture technologies.

Department of Prosthetic Dentistry, Faculty of Dentistry, Ege University , 30 patients who applied for a complete removable denture and met the inclusion criteria will have conventional impressions taken. The resulting master model (reference scan) will be scanned using an industrial scanner with high scanning accuracy (E4 lab scanner, 3shape, Denmark) to obtain digital data. Edentulous ridges; Active Triangulation (Medit i700, Seoul, South Korea), Confocal Microscopy (Trios 5, Henry Schein Dental, Gillingham, Kent, UK), and Multi-Direct-Capture technologies (iTero Lumina, Align Technologies, San Jose, California, USA) will be scanned three times using the scanning protocols recommended by the manufacturers and digitized. All digital data obtained will be evaluated using Geomagic (Studio 2015; 3D Systems Inc., Darmstadt, Germany) 3D analysis software to match the reference data and verify its accuracy according to the accepted reference measurement.

DETAILED DESCRIPTION:
At Ege University Faculty of Dentistry Department of Prosthodontics, Type 4 (hard) plaster will be used to obtain models by taking impressions with Type A silicone impression material from 30 patients undergoing treatment for lower and/or upper complete (total) dentures who meet the inclusion criteria for the study. The model will be scanned using an industrial EOS scanner (E4 lab scanner, 3shape, Denmark). Three digital scans will be taken from each patient using three different IOS scanners (Trios 5 (Henry Schein Dental, Gillingham, Kent, UK), Medit i700 (Seoul, South Korea), and iTero Lumina (Align Technologies, San Jose, California, USA)), with each patient scanned three times using each scanner. The obtained data will be evaluated with a 3D analysis software program (Geomagic Studio 2015; 3D Systems Inc., Darmstadt, Germany) to match the traditional plaster model (reference) data.

For normally distributed data, one-way ANOVA and post hoc Bonferroni test will be performed; for non-normally distributed data, Bonferroni and Kruskal-Wallis tests will be performed. Intergroup comparisons will be tested using the Tukey HSD test. All statistical analyses will be performed using statistical software (IBM SPSS Statistics, v22.0; IBM Corp., USA). It will be investigated whether there is a statistically significant difference in scanning accuracy between the three intraoral scanners.

The study will evaluate three different scanning technologies: Active Triangulation (Medit i700, Seoul, South Korea), Confocal Microscopy technologies (Trios 5, Henry Schein Dental, Gillingham, Kent, UK), and Multi-unit-capture technologies (iTero Lumina, Align Technologies, San Jose, California, USA). A review of the literature reveals that there are few studies evaluating scanners with different technologies in terms of scanning technologies. The aim of this study is to evaluate the accuracy of scanners with different scanning technologies in completely edentulous arches.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 80
* Upper and lower edentulous ridges
* Individuals who have not received radiation therapy or chemotherapy
* Individuals who have not been diagnosed with dry mouth
* Individuals without active mouth sores due to systemic diseases
* Patients who accept the study conditions will be included in the study.

Exclusion Criteria:

* Patients whose extraction site has not yet healed or whose last tooth extraction was less than 2 months ago
* Individuals who have undergone radiation therapy and chemotherapy
* Individuals diagnosed with dry mouth
* Individuals with active mouth sores due to systemic diseases
* Patients who do not agree to the study conditions will not be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Intraoral Scanners Compared With Reference Extraoral Scanner | Two months
  The primary outcome is the trueness (accuracy) of three intraoral scanners (Trios 5, Medit i700, iTero Lumina) in capturing edentulous maxillary and mandibular arches. Accuracy will be assessed by comparing the surface deviation of intraoral scan data to the reference dataset obtained from the extraoral laboratory scanner of a conventional stone cast. Mean root-mean-square (RMS) error values (measured in micrometers, µm) will be calculated for each scanner relative to the reference to quantify the deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University,Faculty of Dentistry,Department of Prosthodontics,Izmir, Izmir, Turkey (Türkiye)